CLINICAL TRIAL: NCT03042949
Title: Correlation of Blood Pressure Measurements Using an Optical System for Measuring Blood Pressure
Brief Title: An Optical System for Measuring Blood Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Naomi Nacasch, Principle Invastigator, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 0265-16-MMC
Record Dates: First submitted 2017-01-31; First posted 2017-02-03 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Blood Pressure Disorders
MeSH Terms: interventions — Blood Pressure Determination

STUDY DESIGN:
Intervention Model Description: Subjects will have their blood pressure measured by standard plethysmography and with a new optical device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood pressure measurement (Experimental): Patients requiring blood pressure measurement will have their blood pressure measured in the standard manner by plethysmography, and then with the Elfor -1 device , the new optical sensor, in order to determine the performance of the new sensor.
  Interventions: Device: Blood pressure measurement; Device: Blood pressure measurement with the new device

INTERVENTIONS:
Device: Blood pressure measurement — Blood pressure measurement with a standard plethysmograph
Device: Blood pressure measurement with the new device — Blood pressure measurement with the optical sensor, Elfor -1 device.

SUMMARY:
An assesment of an optical system that measures blood pressure on the finger -Elfor 1 device. The system is based on a small optical sensor that emits coherent light into the skin and collects the reflected light from the red blood cells in the blood vessels in the skin under the sensor. The sensor is able to detect the pulse wave and blood pressure can be measured.

The investigators plan to measure blood pressure with the new sensor in patients who are attending the Hypertension Clinic at Meir Hospital or are undergoing hemodialysis to validate the sensor.

DETAILED DESCRIPTION:
If the blood flow is temporarily interrupted by inflating a small pneumatic cuff at the root of the finger, blood flow is occluded and the pulse wave disappears. As the pressure in the cuff is released, blood flow returns, the pulse wave is again detected and blood pressure can be measured. This apparatus is easy to use and will allow simplified monitoring of blood pressure contains the laser source and optical sensors that measure the reflected light.

The investigators proposed to validate the sensor by measuring the blood pressure in patients with this optical sensor and also by standard plethysmography. The investigators plan to measure participants with low, normal and high blood pressure in order to assess the accuracy and reliability of the new device.

ELIGIBILITY:
Inclusion Criteria:

* patients on hemodialysis or visiting the hypertension outpatient clinic at Meir Medical Hospital.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-02-15 (Estimated); Primary Completion 2018-02-15 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure reading | three hours
  Measurements will be performed with a standard plethysmograph and with a new sensor

IPD SHARING:
Plan to Share IPD: No